CLINICAL TRIAL: NCT03391037
Title: Internal Jugular Vein Distensibility in Assessment of Fluid Responsiveness in Donors of Living Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Principal investigaror, Ain Shams University
Other Study IDs: 133/2018
Record Dates: First submitted 2017-12-22; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-12

CONDITIONS: Monitoring During Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: diagnostic criteria for volume assessment were heart rate (HR), mean arterial blood pressure (MABP), central venous pressure (CVP), and urine output hourly (UOP) in ml/hr. During period of hypovolemia, all enrolled patients had left IJV scanned (T0) and measured by one anesthesiologist experienced in point-of-care ultrasound. This point-of-care anesthesiologist is not involved in the anesthetic management of the patient and blinded to the volume status of the patient values. Hypovolemic patients were given a fluid bolus in the form of ringer acetate 5 ml / Kg. Ultrasonic and hemodynamic measurements are reassessed 10 minutes (T 10) after the fluid resuscitation.
  Interventions: Diagnostic Test: Internal Jugular Vein Distensibility

INTERVENTIONS:
Diagnostic Test: Internal Jugular Vein Distensibility — . 40 donor candidates for right lobe hepatectomy for living donor liver transplantation were enrolled. During period of hypovolemia (T0) left IJV scanned and measured. After a given fluid bolus in the form of ringer acetate 5 ml / Kg. ultrasonic and hemodynamic measurements were reassessed 10 minutes (T 10) after the fluid resuscitation

SUMMARY:
Egypt has a very high prevalence of HCV and a high morbidity and mortality from chronic liver disease, cirrhosis, and hepatocellular carcinoma. Approximately 20% of Egyptian blood donors are anti-HCV positive. Egypt has higher rates of HCV than neighboring countries as well as other countries in the world with comparable socioeconomic conditions and hygienic standards for invasive medical, dental, or paramedical procedures.

Donor safety is on the top of our priorities as a team and it is widely recognized intraopertively during hepatectomy, there are several potential risks during the Perioperative period .

DETAILED DESCRIPTION:
to a conclusion that intraoperative fluid management aids to the reduction of the intraoperative bleeding during the procedure, adequate and guided fluid management is considered one of the important strategies to reduce the blood loss besides of the other anesthetic techniques like hemodilution, normovolemia, cell salvage usage , high Stroke volume variation (SVV) method ,and low CVP technique , the last method is considered the most applicable, simpler, and cost effective technique which could be easier to be performed.

ELIGIBILITY:
Inclusion Criteria:

* age of 20 years . candidate for donor right lobe hepatectomy for LDLT . volume assessment diagnosed as hypovolemia intraopertively by the anesthesiologist.

Exclusion Criteria:

* inability to scan IJV secondary to surgical dressing, hematoma formation after trial or placement of CVP catheter on left side.

inability for proper positioning.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Prospective blinded observational study
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
correlation between CVP and IJV distensibility | 10 min
  IJV distensibility is the difference between maximum diameter of IJV and minimum diamter in Manchester mode divided by minimum diameter

IPD SHARING:
Plan to Share IPD: Undecided